CLINICAL TRIAL: NCT00039715
Title: Effect of Hydrocortisone Infusion on Hippocampal Glucose Metabolism, Neuropsychological Test Performance and Reexperiencing Symptoms in Patients With Post-Traumatic Stress Disorder (PTSD)
Brief Title: Effects of Hydrocortisone in Patients With Post-Traumatic Stress Disorder
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 020209; 02-M-0209
Record Dates: First submitted 2002-06-06; First posted 2002-06-07 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2004-09

CONDITIONS: Post-Traumatic Stress Disorders; Healthy
Keywords: Glucocorticoid Receptor; Traumatic Reminders; Stress; Hippocampus; Flashbacks; PTSD; Type II GR Receptor; Hydrocortisone; Memory; Major Depression; Post-Traumatic Stress Disorder; Healthy Volunteer; HV; Normal Control
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depressive Disorder, Major

SUMMARY:
The purpose of this study is to determine whether people who develop Post-Traumatic Stress Disorder (PTSD) after a trauma have increased sensitivity to the effects of a stress hormone.

Patients with PTSD have small hippocampal volume and deficits in hippocampal-mediated memory as compared to healthy people. However, it is unclear whether the smaller hippocampi are a consequence of PTSD or a risk factor for the development of PTSD. Some researchers believe that people who develop PTSD have an increase in cortisol levels during traumatic experiences and that this could be neurotoxic to the hippocampus. Others hypothesize that increased sensitivity of glucocorticoid receptors to cortisol, regardless of the cortisol levels, could lead to neurotoxic damage to the hippocampus. This study will compare responses to a stress hormone in patients with PTSD, participants who have experienced trauma but do not have PTSD, and healthy volunteers.

Participants will be screened with a medical and psychiatric interview, physical examination, blood tests, electrocardiogram, and an emotional intelligence evaluation. Those eligible for the study will be asked to collect urine and saliva samples for 3 days. Participation will also include blood draws, a PET scan (brain imaging), an eye-blink test, neuropsychological testing, and other procedures.

At another study visit, participants will undergo a magnetic resonance imaging (MRI) scan (brain imaging), questionnaires, and other procedures.

DETAILED DESCRIPTION:
Patients with post traumatic stress disorder (PTSD) related to combat or civilian trauma have been found to have small hippocampal volume, and deficits in hippocampal mediated memory, compared to the controls. However, it is not clear if the smaller hippocampi are a consequence of the extreme trauma and PTSD, or a risk factor in the development of PTSD. Researchers supporting the causal hypothesis have proposed that increased levels of cortisol during the traumatic experience could be neurotoxic to the hippocampus. Several studies have confirmed an increase in levels of cortisol during stress. However, plasma and urine measures of cortisol in patients with PTSD are mixed; with reports of increased decreased or normal cortisol. The possibility that increased sensitivity of the Type II or glucocorticoid receptors to circulating cortisol could lead to neurotoxic damage to the hippocampus, despite normal to low peripheral levels of cortisol has been proposed. Furthermore, increased sensitivity of the glucocorticoid receptor in PTSD could lead to stronger negative feedback inhibition, thereby offering a mechanism for the paradoxical observation of lower ACTH and cortisol levels in PTSD. Studies attempting to test the glucocorticoid receptor super sensitivity theory in PTSD confirmed the presence of increased number and sensitivity of lymphocyte glucocorticoid receptors in patients compared to healthy subjects. However, there are currently no published reports investigating central glucocorticoid sensitivity in patients with PTSD. A recent study in healthy subjects and Alzheimer's disease demonstrated that central glucocorticoid receptor sensitivity can be measured by hydrocortisone mediated inhibition of glucose metabolism measured by positron emission tomography (PET) and 2-deoxy-2[F]fluoro-D-glucose (FDG). We propose to evaluate the metabolic, cognitive, and behavioral effects of hydrocortisone or placebo administration in patients with PTSD, subjects who have experienced trauma but do not develop PTSD (trauma controls) and healthy subjects.

ELIGIBILITY:
INCLUSION CRITERIA:

1. The study sample will consist of:

   Patients with a primary diagnosis of PTSD due to non-combat or combat related trauma according to DSM-IV.

   Subjects with non-combat related traumatic experiences without current PTSD and

   Healthy subjects without current or past history of psychiatric or major medical illness.
2. All subjects will be between 18 and 60 years old.
3. Male and female subjects will be included.
4. All subjects must be able to give written informed consent prior to participation in this study.
5. Patients with PTSD must score greater than or equal to 50 on Clinician-Administered PTSD Scale as a measure of PTSD symptom severity to be included in the study.
6. Patients who are not currently on medications for PTSD. (Patients will not be discontinued from effective medication for purposes of the study).
7. Patients who are nonresponders to other psychotropic drugs must have discontinued them for at least 2 weeks prior to the first PET scan. Medications will be discontinued under the supervision of the treating physician or a research psychiatrist listed in the protocol. (Nonresponders will be defined as subjects who continue to meet criteria for PTSD despite treatment with 30 mg equivalent of paroxetine for a minimum duration of six weeks).

7. All eligible subjects must be in good physical health as confirmed by a complete physical exam (including normal vital signs), electrocardiogram, neurological exam, and routine laboratory tests of blood and urine. [However, if patients have participated in other research studies or have had blood work through their primary MD within the last 6 months, these results will be used instead of repeating blood draws for inclusion into the study.]

EXCLUSION CRITERIA

1. Subjects with a clinically significant cardiovascular, pulmonary, endocrine, neurological, gastrointestinal illness or unstable medical disorder.
2. Patients who would be unable to comply with study procedures or assessments.
3. Subjects with primary trauma related to motor vehicle accidents.
4. Patients who meet DSM-IV criteria for alcohol and/or substance abuse or substance dependence within 6 months prior to screening.
5. Patients who are currently on fluoxetine (Justification: Washout from fluoxetine could take up to six weeks).
6. Patients who are currently at high risk for homicide or suicide.
7. Subjects with a current or past history of other axis I disorders like schizophrenia, schizoaffective disorder, bipolar disorder or dementia will be excluded from the study. However, those with a comorbid history of other Axis 1 disorder like major depression, dysthymia or panic disorder will be included in the study. Justification: Approximately 70% of subjects with PTSD have comorbid depression and or alcohol abuse; reviewed in 134. Restricting the sample to PTSD patients without depression will not accurately reflect the biology of this disorder].
8. Subjects with a history of peptic ulcer disease will be excluded. (Justification: Those with a history of acid peptic disease requiring antacids in the past will be excluded, although it is unlikely that a single dose of intravenous hydrocortisone could precipitate bleeding due to gastritis or peptic ulcer disease).
9. Women of childbearing potential who are not practicing a clinically accepted method of contraception or who have a positive pregnancy test or who are lactating.
10. Subjects who donated a Red Cross unit of blood within 60 days prior to participation in the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 93
Dates: Start 2002-06; Study Completion 2004-09

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Mental Health (NIMH), Bethesda, Maryland, United States

REFERENCES:
- [Background] Bremner JD, Randall P, Scott TM, Capelli S, Delaney R, McCarthy G, Charney DS. Deficits in short-term memory in adult survivors of childhood abuse. Psychiatry Res. 1995 Nov 29;59(1-2):97-107. doi: 10.1016/0165-1781(95)02800-5. PMID 8771224
- [Background] Bremner JD, Randall P, Scott TM, Bronen RA, Seibyl JP, Southwick SM, Delaney RC, McCarthy G, Charney DS, Innis RB. MRI-based measurement of hippocampal volume in patients with combat-related posttraumatic stress disorder. Am J Psychiatry. 1995 Jul;152(7):973-81. doi: 10.1176/ajp.152.7.973. PMID 7793467
- [Background] Bremner JD, Randall P, Vermetten E, Staib L, Bronen RA, Mazure C, Capelli S, McCarthy G, Innis RB, Charney DS. Magnetic resonance imaging-based measurement of hippocampal volume in posttraumatic stress disorder related to childhood physical and sexual abuse--a preliminary report. Biol Psychiatry. 1997 Jan 1;41(1):23-32. doi: 10.1016/s0006-3223(96)00162-x. PMID 8988792